CLINICAL TRIAL: NCT05879120
Title: Randomized Study of Neo-adjuvant and Adjuvant Pembrolizumab With and Without Targeted Blood Brain Barrier Opening Using Exablate MRI-guided Focused Ultrasound (Exablate MRgFUS) for Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: InSightec (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0812; NCI-2023-04164 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab
- Exablate MRgFUS + neoadjuvant pembolizumab (Experimental)
  Interventions: Device: Exablate MRgFUS + neoadjuvant pembolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: Keytruda; MK-3475; SCH-900475
  Arms: Neoadjuvant pembrolizumab
Device: Exablate MRgFUS + neoadjuvant pembolizumab — Given by IV (vein)
  Arms: Exablate MRgFUS + neoadjuvant pembolizumab

SUMMARY:
To learn if the Exablate Model 4000 Type 2 ("Exablate System") with the DEFINITY® ultrasound contrast agent can temporarily disrupt the blood brain barrier in patients with recurrent (has grown back) glioblastoma who are scheduled to receive pembrolizumab.

DETAILED DESCRIPTION:
Primary Objectives:

1. To estimate the median overall survival (mOS) of BBB opening with neo-adjuvant and adjuvant pembrolizumab and no BBB opening with neo-adjuvant and adjuvant pembrolizumab alone.
2. To assess efficacy of BBB opening with Exablate MRgFUS to enhance intratumoral effector T-cell infiltration during neo-adjuvant and adjuvant pembrolizumab compared to neo-adjuvant and adjuvant pembrolizumab alone.

Secondary Objectives:

1. To characterize safety and describe adverse events associated with opening of the BBB during treatment of recurrent glioblastoma with pembrolizumab.
2. To assess efficacy of BBB opening as measured by drug levels of pembrolizumab in target brain tumor tissue, comparing Exablate MRgFUS BBB opening during neo-adjuvant and adjuvant pembrolizumab compared to neo-adjuvant and adjuvant pembrolizumab alone.
3. To determine anti-tumor activity of pembrolizumab in recurrent glioblastoma, by evaluating PFS, median duration of response, overall response rate, and clinical benefit rate (CR+PR+SD), using modified RANO criteria

Exploratory Objectives:

1. To assess the immunological/biomarker changes, including ctDNA, in peripheral blood and tumor tissue in response to pembrolizumab and MRgFUS in patients with recurrent glioblastoma and to explore any potential association between these biomarker measures and antitumor activity.
2. To determine if neoadjuvant pembrolizumab plus MRgFUS will increases MR contrast enhancement through increased vascular permeability, as well as alter the tumor microenvironment by reducing tumor vascularity, acidity, and hypoxia due to direct anti-tumor activity.
3. To identify alterations in cervical lymph node morphology (size, shape, volume, diffusivity) will correlate with peripheral immune activation and T-cell infiltration into the tumor.
4. To correlate pre-study enrollment MRI tumor growth kinetics with response to treatment.
5. To identify novel immunological correlates of treatment with Pembrolizumab with or without BBB opening with MRgFUS

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of World Health Organization Grade IV glioma (glioblastoma or gliosarcoma) with first recurrence of disease will be enrolled in this study.
2. Only patients with confirmed IDH wild-type glioma will be enrolled in this study.
3. Participants must have undergone prior surgery and completed standard of care treatment with concurrent temozolomide and radiation therapy.
4. Patient is a surgical candidate and resection is indicated as standard of care. Tumor must be supratentorial for surgical candidacy.
5. Surgery is expected to achieve 60% or greater resection of enhancing tumor.
6. A male participant must agree to use a contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 30 days (e.g. 5 terminal half-lives for pembrolizumab and/or any active comparator/combination) plus an additional 90 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period.
7. A female participant is eligible to participate if she is not pregnant (see Appendix 5), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 5 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 5 during the treatment period and for at least 150 days after the last dose of study treatment.
8. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
9. Have unequivocal tumor progression and measurable disease based on mRANO criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
10. Have provided archival tumor tissue sample or biopsy specimen of a tumor not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Receipt of archival tissue is not required for the start of treatment.
11. Have a Karnofsky Performance Score (KPS) of ≥ 70 at the time of enrollment. Evaluaton of KPS is to be performed within 7 days prior to the first dose of study intervention.The participant is on a stable or decreasing dose of steroids of less than or equal to 2 mg dexamethasone per day.
12. Have adequate organ function as defined in the following table (Table 3). Specimens must be collected within 7-14 days prior to the start of study intervention.

    System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1500/µL Platelets ≥100 000/µL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Renal Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR

    ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

    a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

    b Creatinine clearance (CrCl) should be calculated per institutional standard.

    Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
13. All screening labs should be performed with 14 days (+3 working days) of treatment initiation.

    A baseline brain MRI must be obtained no more than 14 days (+3 working days) prior to study enrollment on a stable or tapering dose of steroids no greater than 2 mg a day of dexamethasone (or equivalent) for at least 5 days.
14. For MD Anderson patients only: ability and willingness to consent to protocols PA13-0291 and 2012-0441

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization and each dose of the study treatment. In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of the study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving the study medication. (see Appendix 5). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.
4. Has received prior systemic anti-VEGF or anti-VEGFR treatment (e.g. bevacizumab, cedirinab, aflibercept, vandertanib, XL-184, sunitinib, etc.)
5. Has received prior radiotherapy within 12 weeks of start of study intervention unless there is histologically proven tumor recurrence. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
6. Has received temozolomide within 4 weeks, lomustine within 6 weeks, or any non-cytotoxic tumor directed therapy within 5 half-lives or 2 weeks of start of study intervention.
7. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN] or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
11. Patient's glioblastoma meets criteria to be defined as multifocal or multicentric.
12. Subjects presenting with the following imaging characteristics

    1. Evidence of acute intracranial hemorrhage.
    2. Containing calcifications in the focused ultrasound sonication beam path in the event system tools cannot tailor the treatment around these calcification spots
    3. Evidence of >2 mm midline shift evidence of subfalcine, uncal, or tonsillar herniation on pre-operative imaging
13. The sonication pathway to the tumor involves more than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
14. Ferrous metallic implanted objects in the skull or the brain.
15. Cardiac disease or unstable hemodynamics including:

    1. Documented myocardial infarction within six months of enrollment.
    2. Unstable angina on medication.
    3. Congestive heart failure.
    4. Left ventricular ejection fraction <50%.
    5. History of a hemodynamically unstable cardiac arrhythmia.
    6. Cardiac pacemaker.
16. Stage 2 hypertension defined by the AHA (≥160 systolic or ≥100 mm Hg diastolic on two or more readings (averaged) on two separate occasions) despite standard anti-hypertensive therapy.
17. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment (i.e., antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment).
18. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage
19. Cerebral or systemic vasculopathy, including intracranial thrombosis, vascular malformation, cerebral aneurysm or vasculitis.
20. Evidence of new focal neurological deficits including, but not limited to, motor weakness or speech impairment within 7-14 days prior to the first BBBD procedure.
21. Active drug or alcohol use disorder.
22. Active seizure disorder or epilepsy (seizures despite medical treatment) for a minimum of 4 weeks prior to first cycle/Exablate BBBD procedure captured by history.
23. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
24. Has known active CNS metastases and/or carcinomatous meningitis.
25. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
26. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
27. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/intersitial lung disease.
28. Has active infection requiring systemic therapy within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalizations for complications of infection, bactermia, or severe pneumonia.
29. Signs or symptoms of active infection withn 2 weeks prior to Cycle 1, Day 1
30. Has a known history of Human Immunodeficiency Virus (HIV) infection.
31. Has a known history of active tuberculosis.
32. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HbsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
33. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. Due to the dire nature of the disease for which the research study provides a prospect of direct benefit that is unavailable outside of the trial context, participants with cognitive impairment will be enrolled. Cognitive function will be assessed by treating physician or designee through a neurological examination. The formal consent for such participants will be obtained from their legally authorized representative. However, participants will be informed about the research to the maximum extent compatible with the subject's understanding. Participants will be closely monitored per protocol guidelines and decisions on continuing on study will be based on their treating physician's evaluation of continued benefit or emergence of significant risk. Assent will be obtained from such participants who will sign and date the consent form if capable.
34. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
35. Anticipation of need for a major surgical procedure during the course of the study other than the planned clinical surgery (see Table 1: Schedule of Activities). Definition of what constitutes a major surgical procedure is at the discretion of the site investigator.
36. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
37. Has had an allogenic tissue/solid organ transplant.
38. Contraindication to obtaining MRIs.
39. Known sensitivity to gadolinium-based contrast agents.
40. Known sensitivity to DEFINITY® ultrasound contrast agent.
41. Known hypersensitivity to perflutren microsphere or it components, e.g., polyethylene glycol, as found in Miralax and bowel prep products.
42. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible
43. If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
44. Innability to comply with the study and follow up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Puduvalli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org